CLINICAL TRIAL: NCT03376555
Title: Cheese Consumption and Human Microvascular Function
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lacy Alexander (Other)
Collaborators: National Dairy Council (Other)
Responsible Party: Sponsor-Investigator, Lacy Alexander, Associate Professor of Kinesiology, Penn State University
Organization: Penn State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY4340; 129552 (Other: FDA)
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Microvascular Dysfunction
Keywords: Sodium; Hypertension; Blood Pressure; Cardiovascular Disease; Nitric Oxide; Skin; Dairy; Cheese; Oxidative Stress; Diet; Flow Mediated Vasodilation; Nitroglycerin; Superoxide; Microcirculation
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: All subjects participate in 4 diets in randomized order. The diets differ in the amount of sodium and dairy cheese content. Each diet is consumed for 8 days. Minimum washout of 1 week between diets. Baseline experiment is conducted prior to first dietary intervention, and the experiment is repeated after each dietary intervention.
Masking Description: Investigator and Outcomes Assessor are masked according to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Impact of Dairy and Sodium on Microvascular Health (Experimental): Cross over design with a baseline and 4 dietary interventions
  Interventions: Dietary Supplement: Low sodium no cheese; Dietary Supplement: Low sodium cheese; Dietary Supplement: High sodium no cheese; Dietary Supplement: High sodium cheese

INTERVENTIONS:
Dietary Supplement: Low sodium no cheese — Diet contains 1,500 mg sodium per day Diet does not contain dairy cheese 8 days
Dietary Supplement: Low sodium cheese — Diet contains 1,500 mg sodium per day Diet contains 6 oz dairy cheese per day 8 days
Dietary Supplement: High sodium no cheese — Diet contains 5,500 mg sodium per day Diet does not contain dairy cheese 8 days
Dietary Supplement: High sodium cheese — Diet contains 5,500 mg sodium per day Diet contains 6 oz dairy cheese per day 8 days

SUMMARY:
Increased dairy intake is associated with improved measures of blood vessel health. Dairy cheese, however, is often high in sodium. Dietary sodium can impair blood vessel function. The researchers examine if and how natural cheese may protect against impairments in blood vessel function caused by sodium. For this study, participants complete four 8-day controlled feeding periods in which they eat cheese (6 oz/day) or no cheese during a low-sodium or high-sodium base-diet. The participants complete baseline experiments while on their normal personal diet and then repeat experiments at the end of each controlled feeding period. In some of our experiments, the researchers use a technique called "microdialysis" (MD). With MD, the researchers perfuse some research drugs into the skin on the forearm through tiny tubing that mimics capillaries. These MD drugs mimic or block substances the body naturally makes to control the small blood vessels in the skin. The drugs remain in nickel-sized areas around the tubing and do not go into the rest of the body. The researchers also use a standard technique called "flow mediated dilation" (FMD) that uses blood pressure cuffs and ultrasound to look at the health of larger blood vessels in the body. FMD includes placing a small tablet of nitroglycerin under the tongue during part of the test.

DETAILED DESCRIPTION:
Subject screening will be performed by the Penn State Clinical Translational Research Center (CTRC) medical staff and will include a physical exam by a clinician, anthropometry, and a chemical and lipid profile, liver and renal function. Participants meet with a registered dietitian to determine their caloric energy requirements and identify food preferences. The interview includes surveying the subject's physical activity over the previous 7 days.

Subjects will undergo baseline microdialysis experiments to examine the function of the blood vessels in the skin microcirculation. Subjects will also go through a baseline assessment of conduit vessel endothelial and vascular smooth muscle function with brachial artery flow-mediated vasodilation (FMD), and sublingual nitroglycerin. Following baseline experiments, subjects participate in 4 controlled feeding periods, each 8 days in duration. The controlled feeding periods are assigned in a randomized order. At the end of each 8-day controlled dietary period, subjects will repeat microdialysis experiments, brachial artery FMD, and responsiveness to sublingual nitroglycerin.

ELIGIBILITY:
Inclusion Criteria:

* Seated systolic pressure 120-140 mmHg
* Seated diastolic pressure 70-90 mmHg.
* Normoglycemic (HbA1C <5.7%)

Exclusion Criteria:

* Taking pharmacotherapy that alters peripheral vascular control
* Pregnancy
* Breastfeeding
* Females taking contraceptives (pills, patches, shots, etc.) or hormone replacement therapy
* Taking illicit and/or recreational drugs
* Use of nicotine containing-products (e.g. smoking, chewing tobacco, etc.)
* Known allergy to latex or investigative substances

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lacy M Alexander, PhD, Principal Investigator — Penn State University
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alba BK, Stanhewicz AE, Dey P, Bruno RS, Kenney WL, Alexander LM. Controlled Feeding of an 8-d, High-Dairy Cheese Diet Prevents Sodium-Induced Endothelial Dysfunction in the Cutaneous Microcirculation of Healthy, Older Adults through Reductions in Superoxide. J Nutr. 2020 Jan 1;150(1):55-63. doi: 10.1093/jn/nxz205. PMID 31504721

RESULTS

PARTICIPANT FLOW:
Recruitment Details: July 2017 to October 2019, Centre County, PA
Pre-assignment Details: Subjects were enrolled in 4 separate 8-d controlled feeding interventions in a randomized, crossover study design. All food and beverages were prepared by a registered dietitian in the Pennsylvania State Clinical Research Center Metabolic Kitchen. Investigators involved in data collection and analysis were blinded to the dietary treatment.
Groups:
- Sodium and Dairy Intervention: low sodium no cheese low sodium with cheese high sodium no cheese high sodium with cheese baseline (normal diet)
Period: Overall Study
Arm/Group | Sodium and Dairy Intervention
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Sodium and Dairy Interventions: low sodium no cheese low sodium cheese high sodium no cheese high sodium cheese baseline
Arm/Group | Sodium and Dairy Interventions
Number analyzed (Participants) | 13
Age, Customized [Mean (Standard Deviation); unit: years]
  age | 64 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Microvascular Reactivity to Acetylcholine
Description: Skin blood flow is measured with laser Doppler flowmetry (flux units) and normalized to cutaneous vascular conductance by dividing by mean arterial pressure. Log molar increasing concentrations of acetylcholine are perfused and dose response curves are generated. Dose response curves were analyzed to determine the logEC50 (log Molar)
Time Frame: 1 hour
Population: Data were collected with Windaq (Dataq Instruments) at a frequency of 40 Hz. CVC was calculated as red blood cell flux,. ACh dose concentrations were log-transformed and CVC was expressed as a percentage of maximum. Pharmacological curve modeling was performed using a 4-parameter, nonlinear regression with a variable slope to detect between-diet differences in microvascular sensitivity logEC50 (log Molar) of the group mean curve] to ACh.
Measure: Mean (Standard Error); unit: log (M)
Groups:
- Baseline: Subjects on normal personal diet Acetylcholine (ACh) Dose Response, Local heating (LH), and Flow Mediated Dilation with nitroglycerin experiments
  Acetylcholine (ACh) Dose Response: Probe 1. Lactated Ringer's only (control) Probe 2. Lactated Ringer's + N-G-nitro-L-arginine methyl ester (LNAME) Probe 3. Lactated Ringer's + Ascorbate Probe 4. Lactated Ringer's + Tempol Probe 5. Lactated Ringer's + Apocynin
  Local Heating (LH): Probe 1. Lactated Ringer's only (control) Probe 2. Lactated Ringer's + Ascorbate Probe 3. Lactated Ringer's + Tempol Probe 4. Lactated Ringer's + Apocynin
  Flow Mediated Dilation with nitroglycerin: BP cuff on a forearm, gel on the upper arm just above the elbow, and a Doppler ultrasound probe on the gel. The ultrasound measures vessel size and blood velocity. After a 3-minute "resting" measurement, the cuff inflates for 5 minutes to occlude forearm blood flow (BF). After the cuff deflates, we perform a second reading.
  Sublingual nitroglycerin: The subject is supine. We measure blood pressure. Also, we perform ultrasonography at the brachial artery at the elbow during the procedure. Nurse places a 0.4 mg nitroglycerin tablet under the subject's tongue. The subject remains supine for 20 minutes following the nitroglycerin administration.
- Low Sodium, No Cheese: Diet contains 1,500 mg sodium per day Diet does not contain dairy cheese
  After 8 days on diet:
  Acetylcholine Dose Response, Local heating, and Flow Mediated Dilation with nitroglycerin experiments
  Acetylcholine (ACh) Dose Response: Probe 1. Lactated Ringer's only (control) Probe 2. Lactated Ringer's + N-G-nitro-L-arginine methyl ester (LNAME) Probe 3. Lactated Ringer's + Ascorbate Probe 4. Lactated Ringer's + Tempol Probe 5. Lactated Ringer's + Apocynin
  Local Heating (LH): Probe 1. Lactated Ringer's only (control) Probe 2. Lactated Ringer's + Ascorbate Probe 3. Lactated Ringer's + Tempol Probe 4. Lactated Ringer's + Apocynin
  Flow Mediated Dilation with nitroglycerin: BP cuff on a forearm, gel on the upper arm just above the elbow, and a Doppler ultrasound probe on the gel. The ultrasound measures vessel size and blood velocity. After a 3-minute "resting" measurement, the cuff inflates for 5 minutes to occlude forearm blood flow (BF). After the cuff deflates, we perform a second reading.
  Sublingual nitroglycerin: The subject is supine. We measure blood pressure. Also, we perform ultrasonography at the brachial artery at the elbow during the procedure. Nurse places a 0.4 mg nitroglycerin tablet under the subject's tongue. The subject remains supine for 20 minutes following the nitroglycerin administration.
- Low Sodium, Cheese: Diet contains 1,500 mg sodium per day Diet contains 6 oz dairy cheese per day
  After 8 days on diet:
  Acetylcholine Dose Response, Local heating, and Flow Mediated Dilation with nitroglycerin experiments
  Acetylcholine (ACh) Dose Response: Probe 1. Lactated Ringer's only (control) Probe 2. Lactated Ringer's + N-G-nitro-L-arginine methyl ester (LNAME) Probe 3. Lactated Ringer's + Ascorbate Probe 4. Lactated Ringer's + Tempol Probe 5. Lactated Ringer's + Apocynin
  Local Heating (LH): Probe 1. Lactated Ringer's only (control) Probe 2. Lactated Ringer's + Ascorbate Probe 3. Lactated Ringer's + Tempol Probe 4. Lactated Ringer's + Apocynin
  Flow Mediated Dilation with nitroglycerin: BP cuff on a forearm, gel on the upper arm just above the elbow, and a Doppler ultrasound probe on the gel. The ultrasound measures vessel size and blood velocity. After a 3-minute "resting" measurement, the cuff inflates for 5 minutes to occlude forearm blood flow (BF). After the cuff deflates, we perform a second reading.
  Sublingual nitroglycerin: The subject is supine. We measure blood pressure. Also, we perform ultrasonography at the brachial artery at the elbow during the procedure. Nurse places a 0.4 mg nitroglycerin tablet under the subject's tongue. The subject remains supine for 20 minutes following the nitroglycerin administration.
- High Sodium, No Cheese: Diet contains 5,500 mg sodium per day Diet does not contain dairy cheese
  After 8 days on diet:
  Acetylcholine Dose Response, Local heating, and Flow Mediated Dilation with nitroglycerin experiments
  Acetylcholine (ACh) Dose Response: Probe 1. Lactated Ringer's only (control) Probe 2. Lactated Ringer's + N-G-nitro-L-arginine methyl ester (LNAME) Probe 3. Lactated Ringer's + Ascorbate Probe 4. Lactated Ringer's + Tempol Probe 5. Lactated Ringer's + Apocynin
  Local Heating (LH): Probe 1. Lactated Ringer's only (control) Probe 2. Lactated Ringer's + Ascorbate Probe 3. Lactated Ringer's + Tempol Probe 4. Lactated Ringer's + Apocynin
  Flow Mediated Dilation with nitroglycerin: BP cuff on a forearm, gel on the upper arm just above the elbow, and a Doppler ultrasound probe on the gel. The ultrasound measures vessel size and blood velocity. After a 3-minute "resting" measurement, the cuff inflates for 5 minutes to occlude forearm blood flow (BF). After the cuff deflates, we perform a second reading.
  Sublingual nitroglycerin: The subject is supine. We measure blood pressure. Also, we perform ultrasonography at the brachial artery at the elbow during the procedure. Nurse places a 0.4 mg nitroglycerin tablet under the subject's tongue. The subject remains supine for 20 minutes following the nitroglycerin administration.
- High Sodium, Cheese: Diet contains 5,500 mg sodium per day Diet contains 6 oz dairy cheese per day
  After 8 days on diet:
  Acetylcholine Dose Response, Local heating, and Flow Mediated Dilation with nitroglycerin experiments
  Acetylcholine (ACh) Dose Response: Probe 1. Lactated Ringer's only (control) Probe 2. Lactated Ringer's + N-G-nitro-L-arginine methyl ester (LNAME) Probe 3. Lactated Ringer's + Ascorbate Probe 4. Lactated Ringer's + Tempol Probe 5. Lactated Ringer's + Apocynin
  Local Heating (LH): Probe 1. Lactated Ringer's only (control) Probe 2. Lactated Ringer's + Ascorbate Probe 3. Lactated Ringer's + Tempol Probe 4. Lactated Ringer's + Apocynin
  Flow Mediated Dilation with nitroglycerin: BP cuff on a forearm, gel on the upper arm just above the elbow, and a Doppler ultrasound probe on the gel. The ultrasound measures vessel size and blood velocity. After a 3-minute "resting" measurement, the cuff inflates for 5 minutes to occlude forearm blood flow (BF). After the cuff deflates, we perform a second reading.
  Sublingual nitroglycerin: The subject is supine. We measure blood pressure. Also, we perform ultrasonography at the brachial artery at the elbow during the procedure. Nurse places a 0.4 mg nitroglycerin tablet under the subject's tongue. The subject remains supine for 20 minutes following the nitroglycerin administration.
Arm/Group | Baseline | Low Sodium, No Cheese | Low Sodium, Cheese | High Sodium, No Cheese | High Sodium, Cheese
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11
log (M) | -4.90 (0.2) | -4.82 (0.20) | -5.44 (0.20) | -3.21 (0.55) | -3.21 (0.55)

2. Secondary Outcome: Systolic Blood Pressure
Description: Blood pressure is measured via brachial auscultation manually or with a critical care monitor. The peak blood pressure during a cardiac cycle when the heart contracts.
Time Frame: 8 days
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Baseline | Low Sodium, No Cheese | Low Sodium, Cheese | High Sodium, No Cheese | High Sodium, Cheese
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11
mmHg | 125 (1) | 122 (2) | 121 (3) | 127 (3) | 124 (3)

3. Secondary Outcome: Diastolic Blood Pressure
Description: Blood pressure is measured via brachial auscultation manually or with a critical care monitor. The lowest blood pressure during a cardiac cycle when the heart is between beats.
Time Frame: 8 days
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Baseline | Low Sodium, No Cheese | Low Sodium, Cheese | High Sodium, No Cheese | High Sodium, Cheese
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11
mmHg | 81 (1) | 75 (1) | 74 (1) | 78 (1) | 76 (1)

4. Secondary Outcome: Flow Mediated Dilation
Description: Flow mediated dilation is measured through Doppler ultrasound probe placed at brachial artery.
Time Frame: 8 days
Measure: Mean (Standard Error); unit: percentage of flow mediated vasodilation
Arm/Group | Baseline | Low Sodium, No Cheese | Low Sodium, Cheese | High Sodium, No Cheese | High Sodium, Cheese
Number analyzed (Participants) | 7 | 9 | 8 | 7 | 5
percentage of flow mediated vasodilation | 3.78 (0.78) | 5.07 (0.90) | 4.20 (0.76) | 3.45 (1.04) | 5.90 (1.34)

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Baseline | Low Sodium, No Cheese | Low Sodium, Cheese | High Sodium, No Cheese | High Sodium, Cheese
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT03376555/Prot_SAP_ICF_000.pdf